CLINICAL TRIAL: NCT01262183
Title: A Randomised Phase II Study of Radio-chemotherapy With or Without Panitumumab (Vectibix®) in Irresectable Squamous Cell Carcinoma or Adenocarcinoma of the Oesophagus
Brief Title: Radio-chemotherapy With or Without Panitumumab (Vectibix®) in Irresectable Squamous Cell Carcinoma or Adenocarcinoma of the Oesophagus
Acronym: PANORAMIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment numbers
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO200905
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-04

CONDITIONS: Irresectable Squamous Cell or Adenocarcinoma of the Oesophagus
Keywords: oesophagus cancer; chemoradiotherapy; panitumumab; irresectable
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiation therapy with panitumumab (Experimental)
  Interventions: Drug: CRT + Panitumumab
- Concurrent chemoradiation therapy without panitumumab (Active Comparator)
  Interventions: Drug: Concurrent chemoradiation therapy without panitumumab

INTERVENTIONS:
Drug: CRT + Panitumumab — Day -7, day +15 and day +36: panitumumab 9.0 mg/kg i.v. Day +1 to +39: radiation therapy 1.8 Gy fractions 5 times per week to a cumulative dose of 50.4 Gy Day +1 and +29: cisplatin 75 mg/m2 i.v. Day +1 to +4 and +29 to +32: 5-fluorouracil 1000 mg/m2 i.v.
  Arms: Concurrent chemoradiation therapy with panitumumab
Drug: Concurrent chemoradiation therapy without panitumumab — Day +1 to +39: radiation therapy 1.8 Gy fractions 5 times per week to a cumulative dose of 50.4 Gy Day +1 and +29: cisplatin 75 mg/m2 i.v. Day +1 to +4 and +29 to +32: 5-fluorouracil 1000 mg/m2 i.v.
  Arms: Concurrent chemoradiation therapy without panitumumab

SUMMARY:
For esophageal cancer that can not be removed by surgery, the choice of treatment is a combination of chemotherapy and radiotherapy. We call this combination- (or concurrent) chemoradiotherapy. Chemotherapy is treatment with drugs that kill cancer cells. Both chemotherapy and radiotherapy make the tumour smaller and enhance each other's effect. The goal of treatment with chemotherapy and radiation therapy is to cure the cancer. Unfortunately only a small proportion of patients are cured with this treatment.

Improvements in the outcome of treatment may be expected by using the so-called "targeted" treatments. With esophageal cancer, a protein (the epidermal growth factor receptor (this is a kind of trap), the EGFR), is present in many tumours. This protein causes the tumor to grow. Panitumumab is a drug that blocks the functioning of this receptor (catcher), so that possibly the growth and spread of esophageal cancer is prevented.

The main objective of this trial is to see if survival of patients with inoperable esophageal cancer improves as panitumumab is added to standard treatment with chemoradiotherapy.

It will also investigate whether patients tolerate the addition of panitumumab to the standard treatment. Also, the biological characteristics of the tumor will be examined. In a proportion of patients it will be determined how the enhancement of the cancer is visible on an FDG-PET scan before the start of treatment and how this changes during the treatment. It will be also be evaluated how this treatment affects the survival.

DETAILED DESCRIPTION:
A complete response rate of approximately 30% is achieved for standard treatment of irresectable carcinoma of the oesophagus, consisting of concurrent chemoradiation therapy (50.5 Gy + cisplatin/5-FU). Attempts to improve outcome by intensifying conventional cytotoxic drugs or increasing the radiation dose have not been successful. Future improvements will likely require the incorporation of targeted agents that probably will not add significant toxicity, the use of molecular predictors of response and early identification of responders. In both squamous cell carcinoma and adenocarcinoma of the oesophagus expression of EGFR is correlated with poor outcome. Furthermore the addition of cetuximab, a chimaeric EGFR antibody, to radiation therapy in head and neck cancer and non-small cell lung cancer showed a gain in overall survival. In head and neck cancer studies with the addition of panitumumab to chemo-radiation therapy are currently ongoing. Therefore, we propose to perform a randomised phase II study of chemo-radiation therapy with or without the combination of panitumumab (human EGFR antibody) in irresectable squamous cell carcinoma or adenocarcinoma of the oesophagus without distant metastases.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70years
* Histology proven SCC or adenocarcinoma of the oesophagus
* No proven (distant) metastases (ultrasonography, CT or MRI)
* No prior treatment for carcinoma of the oesophagus
* Karnofsky performance status ≥70% (appendix A)
* Irresectable disease as assessed by the multidisciplinary tumour board
* All patients (male and female) must use effective contraception methods according to CPMP/ICH/286/95 if of reproductive potential (e.g. implants, injectables, combined oral contraceptives, IUDs, sexual abstinence or vasectomised partner), for the whole duration of the study and until six months after they received the last treatment dose
* No contraindications for cytotoxic therapy or panitumumab:
* No known hypersensitivity/allergy to any of the compounds used
* Haematology: Neutrophil count ≥ 1.5∙109 /L Thrombocyte count ≥ 100∙109 /L Haemoglobin ≥ 6.2 mmol/L (100 g/L)
* No known HIV infection or other condition of persistent immunodeficiency
* Renal function:
* Creatinine clearance (MDRD) ≥ 60 mL/min
* Hepatic function:
* Total bilirubin ≤ 1.5∙ULN
* AST, ALT, AP ≤ 2.5∙ULN
* Electrolyte balance:
* (albumin corrected) calcium ≤ 2.87 mmol/L (=11.5 mg/dl) but ≥ lower limit of normal (LLN)
* Magnesium ≥ LLN
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* No known other serious illness or medical condition present at entry in the study including: Unstable cardiac disease despite treatment, congestive heart failure NYHA grade 3 and 4 Clinically significantly abnormal electrocardiogram (ECG) or left ventricular ejection fraction (LVEF) below the institutional ULN
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment/randomisation
* Significant neurologic or psychiatric disorders
* Active uncontrolled infection Active disseminated intravasal coagulation
* Symptomatic peripheral neuropathy (CTCAE v3.0 term "neuropathy: sensory") ≥ grade 2 Ototoxicity (CTCAE v3.0 any term in "auditory/ear") ≥ grade 2 except if due to trauma or mechanical impairment due to tumour mass
* Other serious underlying medical condition which could impair the ability of the patient to participate in the study No or insufficient oral nutrient intake
* No prior exposure to EGFR pathway targeting agents
* No known drug abuse
* Absence of any psychological, familial, sociological (e.g. severe alcohol addiction expected to hamper protocol compliance) or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* No participation in another interventional clinical trial in the preceding 30 days
* Written informed consent to participate to study must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Prior treatment for this tumour
* Prior treatment with radiation therapy in the area of the oesophagus or other site that will interfere with proposed treatment
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
* History of other prior malignancy in past 5 years, other than basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.

Exclusion criteria for the PET-scan (secondary endpoint)

For the PET-scan the following exclusion criteria are used:

* Severe claustrophobia
* Diabetes mellitus (type I and II)
* Serum glucose level >11 mmol/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
1-year overall survival | 1-year
  To describe the 1-year OS rate after concurrent CRT with or without panitumumab in irresectable carcinoma of the oesophagus. The control arm is used to validate whether the historical cohort used for comparison is similar to our success-rate.

SECONDARY OUTCOMES:
toxicity | during treatment and follow up
  Investigation of the acute and long-term toxicity of both study arms (according to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0);
PFS | between randomisation and date of PD
  PFS: interval between randomisation date and the date at which disease progression is established being not suspicious for a second cancer (histologically confirmed when in doubt) or date of death from any cause but clearly not related to disease- or treatment (e.g. accident). Patients still disease-free after 18 months follow-up or lost to follow-up or death clearly not related to disease or treatment (e.g. accident)), are censored at the date of the most recent follow-up or at the analysis cut-off date, whichever comes first.
Response Rate | 3 months after treatment
  Response rate: partial (PR) or complete response (CR) according to RECIST 1.1 at 3 months after treatment
pharmacodynamics of panitumumab | biopsy at baseline (standard) and the biopsy one week after start chemo-radiation therapy
  pharmacodynamics (PD) of panitumumab (EGFR, K-RAS, B-RAF, downstream signalling pathways ) compared between the biopsy at baseline (standard) and the biopsy one week after start chemo-radiation therapy
Quantification of baseline FDG uptake (SUV) with PET, and SUV changes | baseline 7 days after the first panitumumab dose or for start chemo-radiation therapy. during treatment with chemoradiation therapy after three weeks.
  baseline, 7 days after the first panitumumab dose or for start chemo-radiation therapy. during treatment with chemoradiation therapy after three weeks.
  2-4 weeks after finishing treatment. 10-12 weeks after finishing treatment
CTCs and CECs | baseline,after 2 weeks during chemo-radiation therapy and 12 weeks after finishing treatment

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, Md PhD, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Gelderland, Netherlands